CLINICAL TRIAL: NCT04062526
Title: Evaluation of in Vivo Neuroinflammation in Parkinson's Disease Using 18F-NOS Positron Emission Tomography (PET/CT)
Brief Title: Evaluation of Neuroinflammation in Parkinson's Disease Using 18F-NOS PET/CT
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 833589
Record Dates: First submitted 2019-08-14; First posted 2019-08-20 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Parkinson Disease; Healthy Volunteer
MeSH Terms: conditions — Parkinson Disease | interventions — Fluorine-18

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Patient with Parkinson Disease (Experimental): Subject should have a history of diagnosis of probable idiopathic PD derived from UK Brain Bank Diagnostic criteria per neurologist review.
  Subject must have been diagnosed with Parkinson's Disease at least 3 year prior to enrollment.
  Interventions: Drug: [18F]NOS
- Healthy Control (Experimental): Subject must be a Healthy.
  Interventions: Drug: [18F]NOS

INTERVENTIONS:
Drug: [18F]NOS — [18F]NOS is an investigational radiotracer which each subject will have one [18F]NOS positron emission tomography/computed tomography (PET/CT) scan performed.
  Other Names: [18F]-6-(2-fluoro-propyl)-4-methylpyridin-2-amine

SUMMARY:
The research study is being conducted to test how a specialized type of Positron Emission Tomography (PET/CT) scan could potentially be useful in diagnosing or monitoring treatment in people with Parkinson's disease. If the subject decide to be in this study he/she will have a PET/CT scans using an imaging drug called 18F-NOS which will be used to measure inflammation in the brain.

DETAILED DESCRIPTION:
The purpose of this research is to test whether it is possible to measure inflammation in subject's brain using an imaging scan called Positron Emission Tomography / Computed Tomography (PET/CT). There are two groups of people who will participate in this study, a Parkinson's disease (PD) group and a Control group Both groups will have imaging with a radioactive drug called 18F-NOS which is an experimental radioactive drug used in PET/CT imaging to measure inflammation in the brain. 18F-NOS has not yet been approved by the Food and Drug Administration (FDA) for use except in a research study. The use 18F-NOS in this study is allowed under an Investigational New Drug Application approved by the FDA.

If subject agree to participate in this study, she/ he will undergo one experimental 18F-NOS PET/CT scan. During the scan, PET/CT images will be taken of subject head in order to capture pictures of their brain. The imaging procedures will be explained to subject in more detail below. Blood samples will be taken at various time points to measure the concentration of the imaging drug in your blood during the scan and a blood sample will be collected to measure specialized inflammation markers in the blood.

Investigator hopes to compare the PET/CT scans for the two groups to see if there are differences between Parkinson patients and Controls. Investigator will also compare the results with other informationgathered about subject during their participation, including brain MRI and inflammation markers.

ELIGIBILITY:
Inclusion Criteria (HC and PD cohorts)

1. Participants will be 18-75 years of age.
2. Participants must be informed of the investigational nature of this study and be willing to provide written informed consent and participate in this study in accordance with institutional and federal guidelines prior to study-specific procedures.
3. Subjects with known neuropsychiatric disorder may be eligible if, in the opinion of an investigator, the psychiatric condition would not compromise subject safety or successful participation in the study.

Inclusion Criteria (PD cohort only)

1. History of diagnosis of probable idiopathic PD derived from UK Brain Bank Diagnostic criteria(1) per neurologist review.
2. Diagnosed with Parkinson's Disease at least 3 year prior to enrollment.
3. Subjects will be selected who have the capacity to give their own informed consent, in the opinion of a neurology investigator.

Exclusion Criteria (HC and PD cohorts)

1. Females who are pregnant or breast feeding at the time of screening will not be eligible for this study; a urine pregnancy test will be performed in women of child- bearing potential within one day of the PET/CT scan.
2. At screening, the participant's weight is > 350 lb.
3. Subject reported claustrophobia that in the opinion of an investigator would interfere with acquisition of the structural MRI required for PET co-registration, and/or the PET scan itself.
4. History of epilepsy or seizure disorder as assessed by medical record review and/or self-report.
5. History of head trauma that in the opinion of an investigator may interfere with the uptake of applicable radiotracer as assessed by medical record review and/or self- report.
6. Current tobacco or nicotine dependence. History of greater than 5 pack years of smoking and less than 2 years since smoking cessation.
7. Self-reported current alcohol consumption of greater than or equal to 25 drinks per week.
8. Inability to tolerate imaging procedures in the opinion of an investigator or treating physician.
9. Any current medical condition, illness, or disorder as assessed by medical record review and/or self-reported that is considered by a physician or investigator to be a condition that could compromise participant safety or successful participation in the study.

Exclusion Criteria (HC cohort only)

1. History of first degree relative with Parkinson's Disease.
2. Use of a CNS drug (prescription, over-the counter or recreational) within 30 days of screening, as assessed by review of medical history and concomitant medication review at screening (from medical record and/or self-report) that are deemed by a physician or investigator to have a potential influence on the binding of the applicable radiotracer.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-08-14 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Characterize the uptake of [18F]NOS | 3 years
  Characterize the uptake of [18F]NOS in the human brain for healthy controls and PD patients.

SECONDARY OUTCOMES:
Compare patterns of uptake | 3 years
  Compare patterns of [18F]NOS brain uptake in patients with PD versus healthy controls.
Compare peripheral blood inflammatory biomarkers | 3 years
  Compare peripheral blood inflammatory biomarkers, including cytokines and mtDAMPs, in PD patients with healthy controls.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Dubroff, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States